CLINICAL TRIAL: NCT00332254
Title: IL-1ra for Prevention of Chondropathy Following Knee Injury
Brief Title: Study to Prevent Cartilage Damage Following Acute Knee Injury.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00014439; 7939-05-11 (Other: Duke IRB#)
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2008-01

CONDITIONS: Knee Injury
Keywords: Anterior cruciate ligament tear; Meniscus tear; Chondral injury
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intra-articular IL-1Ra
  Interventions: Drug: Anakinra
- 2 (Placebo Comparator): Intra-articular saline
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 150 mg IL1Ra ia x1 vs saline ia x1
  Other Names: Kineret

SUMMARY:
Individuals who have had a severe knee injury have an increased risk of developing arthritis of the knee and at a much earlier age than would otherwise be expected. The swelling and inflammation that occur after injury are believed to be responsible for this cartilage damage. The cartilage (material that provides a cushion in the knee) is the primary protection from what is called degenerative arthritis or osteoarthritis. We hope to reduce this swelling and prevent the damage to cartilage that occurs after injury by injecting a medication that blocks one of the proteins responsible for inflammation and cartilage breakdown. This protein is called interleukin-1 and can be inhibited by an interleukin-1 receptor antagonist called anakinra. Anakinra will be injected directly into the injured knee and response to the injection will be measured by symptoms and analysis of cartilage breakdown in the knee fluid and blood.

DETAILED DESCRIPTION:
Osteoarthritis is highly prevalent with significant impact on health care utilization and personal suffering. Injury predisposes to OA even after surgical correction (1, 2). Definitive therapy for established OA is lacking and current treatments are increasingly questioned with regard to long-term safety. Interleukin-1 is instrumental in OA pathogenesis (3-5). Recent studies by Chevalier demonstrated that intra-articular use of IL-1ra was safe in patients with established OA (6). We hope to show that IL-1ra will provide symptomatic benefit after knee injury as well as decreasing cartilage breakdown.

The trial will consist of trial administering 150mg of Anakinra, or placebo, within 30 days of an acute knee injury that requires surgical repair. We hypothesize that higher IL-1 in synovial fluid after injury will predict greater symptomatic response to IL-1ra. Outcome measures will be functional and pain assessments at regular intervals before and after surgery (7, 8). Cartilage catabolism will be assessed with two primary measures. First we will assess degree of chondropathy via direct cartilage visualization and scoring at the time of arthroscopic repair (9). Secondly, the impact of IL-1ra on the inflammatory milieu will be determined through analysis of serum and synovial fluid cytokine levels and cartilage biomarkers at enrollment and again at the time of surgical repair.

The impetus for this study is based on previous work done in animal models of OA, showing prevention of cartilage damage following surgically induced ACL injury (10-12). We believe that intra-articular delivery of anakinra within a short time following knee injury will improve patient function and pain reporting and will also prevent chondropathy that results from injury.

ELIGIBILITY:
Inclusion Criteria:

* Onset of injury less than 4 weeks prior to evaluation
* Severe knee injury that requires surgery, including anterior cruciate ligament tear, meniscus tear and chondral injury
* BMI less than 30
* Age 18-30
* Women will have serum pregnancy testing (bHCG) at time of entry and on follow-up evaluation and must agree to use an approved form of contraception during the study period.

Exclusion Criteria:

* Prior signal joint injury requiring medical evaluation
* History of arthritis or rheumatic disease
* History of intra-articular corticosteroid in index joint
* Septic joint
* Evidence of chronic joint disease by plain radiograph
* Fracture or multiple ligament tear
* Pregnancy or lactation
* Inability to give informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
pain | 4 and 30 days

SECONDARY OUTCOMES:
chondropathy score | 30-60 days

CONTACTS AND LOCATIONS:
Overall Officials: Virginia B Kraus, MD, PhD, Study Chair — Duke University
Locations (1):
- Duke University Sports Medicine Clinic, Durham, North Carolina, United States

REFERENCES:
- [Background] Gelber AC, Hochberg MC, Mead LA, Wang NY, Wigley FM, Klag MJ. Joint injury in young adults and risk for subsequent knee and hip osteoarthritis. Ann Intern Med. 2000 Sep 5;133(5):321-8. doi: 10.7326/0003-4819-133-5-200009050-00007. PMID 10979876
- [Background] Roos EM. Joint injury causes knee osteoarthritis in young adults. Curr Opin Rheumatol. 2005 Mar;17(2):195-200. doi: 10.1097/01.bor.0000151406.64393.00. PMID 15711235
- [Background] Pelletier JP, DiBattista JA, Roughley P, McCollum R, Martel-Pelletier J. Cytokines and inflammation in cartilage degradation. Rheum Dis Clin North Am. 1993 Aug;19(3):545-68. PMID 8210574
- [Background] Pelletier JP, McCollum R, Cloutier JM, Martel-Pelletier J. Synthesis of metalloproteases and interleukin 6 (IL-6) in human osteoarthritic synovial membrane is an IL-1 mediated process. J Rheumatol Suppl. 1995 Feb;43:109-14. PMID 7752112
- [Background] Lotz M. Cytokines in cartilage injury and repair. Clin Orthop Relat Res. 2001 Oct;(391 Suppl):S108-15. doi: 10.1097/00003086-200110001-00011. PMID 11603695
- [Background] Chevalier X, Giraudeau B, Conrozier T, Marliere J, Kiefer P, Goupille P. Safety study of intraarticular injection of interleukin 1 receptor antagonist in patients with painful knee osteoarthritis: a multicenter study. J Rheumatol. 2005 Jul;32(7):1317-23. PMID 15996071
- [Background] Paxton EW, Fithian DC, Stone ML, Silva P. The reliability and validity of knee-specific and general health instruments in assessing acute patellar dislocation outcomes. Am J Sports Med. 2003 Jul-Aug;31(4):487-92. doi: 10.1177/03635465030310040201. PMID 12860533
- [Background] Irrgang JJ, Anderson AF. Development and validation of health-related quality of life measures for the knee. Clin Orthop Relat Res. 2002 Sep;(402):95-109. doi: 10.1097/00003086-200209000-00009. PMID 12218475
- [Background] Ayral X, Dougados M, Listrat V, Bonvarlet JP, Simonnet J, Poiraudeau S, Amor B. Chondroscopy: a new method for scoring chondropathy. Semin Arthritis Rheum. 1993 Apr;22(5):289-97. doi: 10.1016/s0049-0172(05)80008-3. PMID 8511593
- [Background] Pelletier JP, Caron JP, Evans C, Robbins PD, Georgescu HI, Jovanovic D, Fernandes JC, Martel-Pelletier J. In vivo suppression of early experimental osteoarthritis by interleukin-1 receptor antagonist using gene therapy. Arthritis Rheum. 1997 Jun;40(6):1012-9. doi: 10.1002/art.1780400604. PMID 9182910
- [Background] Fernandes J, Tardif G, Martel-Pelletier J, Lascau-Coman V, Dupuis M, Moldovan F, Sheppard M, Krishnan BR, Pelletier JP. In vivo transfer of interleukin-1 receptor antagonist gene in osteoarthritic rabbit knee joints: prevention of osteoarthritis progression. Am J Pathol. 1999 Apr;154(4):1159-69. doi: 10.1016/S0002-9440(10)65368-0. PMID 10233854
- [Background] Caron JP, Fernandes JC, Martel-Pelletier J, Tardif G, Mineau F, Geng C, Pelletier JP. Chondroprotective effect of intraarticular injections of interleukin-1 receptor antagonist in experimental osteoarthritis. Suppression of collagenase-1 expression. Arthritis Rheum. 1996 Sep;39(9):1535-44. doi: 10.1002/art.1780390914. PMID 8814066
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Kessler S, Lang S, Puhl W, Stove J. [The Knee Injury and Osteoarthritis Outcome Score--a multifunctional questionnaire to measure outcome in knee arthroplasty]. Z Orthop Ihre Grenzgeb. 2003 May-Jun;141(3):277-82. doi: 10.1055/s-2003-40083. German. PMID 12822074
- [Background] Marks PH, Donaldson ML. Inflammatory cytokine profiles associated with chondral damage in the anterior cruciate ligament-deficient knee. Arthroscopy. 2005 Nov;21(11):1342-7. doi: 10.1016/j.arthro.2005.08.034. PMID 16325085
- [Background] Poole AR, Ionescu M, Fitzcharles MA, Billinghurst RC. The assessment of cartilage degradation in vivo: development of an immunoassay for the measurement in body fluids of type II collagen cleaved by collagenases. J Immunol Methods. 2004 Nov;294(1-2):145-53. doi: 10.1016/j.jim.2004.09.005. PMID 15637808
- [Background] Matyas JR, Atley L, Ionescu M, Eyre DR, Poole AR. Analysis of cartilage biomarkers in the early phases of canine experimental osteoarthritis. Arthritis Rheum. 2004 Feb;50(2):543-52. doi: 10.1002/art.20027. PMID 14872497
- [Derived] Kraus VB, Birmingham J, Stabler TV, Feng S, Taylor DC, Moorman CT 3rd, Garrett WE, Toth AP. Effects of intraarticular IL1-Ra for acute anterior cruciate ligament knee injury: a randomized controlled pilot trial (NCT00332254). Osteoarthritis Cartilage. 2012 Apr;20(4):271-8. doi: 10.1016/j.joca.2011.12.009. Epub 2012 Jan 10. PMID 22273632
- [Derived] Catterall JB, Stabler TV, Flannery CR, Kraus VB. Changes in serum and synovial fluid biomarkers after acute injury (NCT00332254). Arthritis Res Ther. 2010;12(6):R229. doi: 10.1186/ar3216. Epub 2010 Dec 31. PMID 21194441